CLINICAL TRIAL: NCT06982339
Title: Beat the Heat: Impacts of Heat on Health in Boston and Strategies to Address Them
Brief Title: Beat the Heat Boston
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Gary Adamkiewicz, Associate Professor of Environmental Health and Exposure Disparities, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB25-0366; 1P20TW013028-01 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-08

CONDITIONS: Hot Weather; Adverse Effect; Heat Effect; Heat Stress; Heat Stroke, Heat Exhaustion; Heat Exposure; Heat Strain
Keywords: Cooling; Air conditioner; Heat related illness; stepped wedge
MeSH Terms: conditions — Heat Stress Disorders; Heat Stroke; Heat Exhaustion

STUDY DESIGN:
Intervention Model Description: This study follows a stepped wedge randomized controlled trial (SW-RCT) design to evaluate the health and environmental impacts of air conditioning among older adults with chronic health conditions. A total of 100 participants are randomized into two groups:
  Arm A (Early AC Group): Receives a window AC unit in Year 1, along with a financial subsidy for electricity..
  Arm B (Delayed AC Group): Receives an identical AC unit in Year 2, along with a financial subsidy for electricity.
  In Year 1, participants in Arm A (AC) are compared to those in Arm B (no AC) to assess the direct effect of AC access.
  In Year 2, both arms have AC units, but only Arm B receives the electricity subsidy, allowing evaluation of cost as a barrier to use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Air Conditioning (Experimental): Year 1: Participants receive a window AC unit and a financial subsidy for electricity.
  Year 2: Participants continue to have their AC unit, but do not receive a financial subsidy for electricity.
  Interventions: Other: Air Conditioner; Other: Electricity subsidy
- Delayed Air Conditioning (No Intervention): Year 1: No intervention. Year 2: Participants receive an AC unit along with a financial subsidy for electricity.

INTERVENTIONS:
Other: Air Conditioner — Air conditioners will be window-mounted units powered by 110v AC.
  Arms: Early Air Conditioning
Other: Electricity subsidy — Electricity subsidies will consist of a single block subsidy of USD 100, intended to provide support for the electricity costs associated with operating an air conditioning unit.
  Arms: Early Air Conditioning

SUMMARY:
The goal of this stepped wedge trial is to assess the practical effects of air conditioners on hot weather impacts among older adults. The main questions it aims to answer are:

How does the presence of an air conditioning unit affect heat stress, heat strain, mental health, and healthcare utilization among older adults who did not previously have access to air conditioning?

How, and in what conditioners, do older adults use air conditioning once it is installed in their home?

Researchers will compare participants in arms with (A) and without (B) air conditioning units in the first summer season; this will allow them to assess the effect of air conditioners. In the second summer season, both arms will have air conditioning units, but those in the year two distribution arm (B) will receive an electricity subsidy, while those in the year one AC distribution arm (A) will not, allowing researchers to assess the effect of an electricity subsidy.

Participants will be randomized to receive an air conditioner and financial support for electricity costs in either the first summer season or the second summer season of the study.

* Heat stress, heat strain, mental health, and healthcare utilization will be assessed via participant survey.
* Air conditioner utilization will be assessed via continuous load monitoring devices.
* Indoor air temperature will be assessed via continuous data loggers.

DETAILED DESCRIPTION:
This community-based, randomized stepped wedge trial investigates whether the provision of educational resources and air conditioning (AC) improves thermal comfort and health outcomes among older adults with chronic disease and material hardships. The study will enroll 100 participants residing in at risk neighborhoods. Eligibility criteria include adults aged 55-95 who speak English or Spanish, lack access to home cooling systems, and have at least one qualifying chronic health condition or a history of recent hospitalization (see Eligibility section) .

Participants will be randomly assigned (1:1) to receive window AC units and an electricity cost subsidy either in Year 1 or Year 2. All participants in both arms will receive a baseline intervention including heat health educational materials and cooling kits. Data collection will occur over two warm seasons (April-September) and involve pre- and post-intervention assessments using structured surveys, real-time environmental monitoring, and AC usage tracking.

Surveys administered at enrollment and in late summer each year will capture a broad range of covariates including sociodemographic data, housing conditions, health service utilization, self-reported symptoms, and adaptive behaviors. Heat stress, heat strain, mental health, and healthcare utilization outcomes will be assessed via surveys that include previously validated survey instruments. Specific emphasis will be placed on measures of energy insecurity, such as utility shutoff notices, receipt of energy assistance, and trade-offs between essential expenses. Environmental sensors will log indoor temperature, humidity, and pollutant data throughout the study period.

The primary outcome is self-reported health status as measured by a modified ESQ-IV, supplemented by secondary metrics including ASHRAE thermal comfort scores, POMS, emergency department presentations, and hospitalizations. Statistical analysis will employ two-sample t-tests to detect treatment effects, with a minimum detectable effect size of 5.66 assuming a standard deviation of 10 and balanced sample sizes.

This study aims to empirically quantify the health benefits of cooling interventions in high-risk older adults and inform scalable public health strategies that address the intersecting challenges of urban heat, chronic disease management, and housing-related inequities.

ELIGIBILITY:
Inclusion Criteria:

* reside in Roxbury, Dorchester, East Boston or Mattapan MA
* age 55-95 years old
* speak English or Spanish
* do not have air conditioning in the home
* living with at least one of the following conditions: chronic CVD (hypertension, hyperlipidemia, diabetes, history of stroke or myocardial infarction, atrial fibrillation, or heart failure), chronic pulmonary disease (asthma, COPD/emphysema, interstitial lung disease), chronic neurologic disease (stroke, Parkinson's disease, or other chronic neurologic conditions), chronic mental health conditions (including anxiety disorder, major depression, bipolar disorder), and/or history of hospitalization (defined as spending at least one night in the hospital) for any reason within the past three years.

Exclusion Criteria:

- Lack a location in their home suitable for installation of the AC unit provided during the research study.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Environmental Symptoms Questionnaire (ESQ-IV) | Difference in self-reported symptoms on HSSQ administered in the late summer season, 2-12 weeks after enrollment.
  The primary outcome will be a two-sample t-test for differences in means in the treatment and control groups in responses to the Environmental Symptoms Questionnaire (ESQ-IV).
  We will assess self-reported health impacts across all sites using a modified (truncated) version of the Environmental Symptoms Questionnaire (ESQ-IV), referred to as the Heat Stress Symptoms Questionnaire. Originally developed for assessing the health impacts of environmental exposures (Sampson et al, 1993), the ESQ-IV has been validated for assessing health impacts associated with heat illness in soldiers (Johnson & Merullo, 1993). More recently, smaller subsets of the ESQ-IV's questions have served as a health endpoint for assessing the impacts of heat stress and acclimatization in the general population and older adults (McGarr et al, 2023; Manning et al, 2023). In an urban population, a question using similar language in a simplified format was used to assess prior experiences of heat-related illness (Card

SECONDARY OUTCOMES:
Air Conditioner Utilization | From enrollment to study completion, approximately 2 years.
  Air conditioner utilization will be prospectively assessed throughout the study. In year 1, air conditioner utilization will be analyzed in relation to indoor air temperature to identify threshold temperatures that trigger AC utilization. In Year 2, utilization rates and thresholds will be compared between the the two arms to assess the impact of electricity subsidies on AC utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Adamkiewicz Associate Professor of Environmental Health and Exposure Disp., PhD, MPH, MS, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable study dataset, specifically data on treatment arm assignment and survey results including primary endpoint
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of publication of study results.
Access Criteria: Data will be available upon reasonable request.